CLINICAL TRIAL: NCT04580355
Title: Impact of Non-surgical Periodontal Therapy With or Without Antibiotics on Oral and Gut Microbiome in Patients With Stage III/IV and Grade C Periodontitis
Brief Title: Impact of Non-surgical Periodontal Therapy on Oral and Gut Microbiome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Professor of Periodontics in Piracicaba Dental School-FOP/UNICAMP, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23626219.7.0000.5418
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Microbial Colonization; Periodontal Diseases; Periodontal Inflammation
MeSH Terms: conditions — Communicable Diseases; Periodontal Diseases | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMUD + Placebos (Experimental): One session of full-mouth ultrasonic debridement (FMUD) with a time limit of 45 minutes plus placebo administration prescribed on the day of treatment, every 8 hours for 7 days.
  Interventions: Procedure: One-Stage Full Mouth Debridement; Drug: Amoxicillin Placebo; Drug: Metronidazole Placebo
- FMUD + AM (Active Comparator): One session of full-mouth ultrasonic debridement (FMUD) with a time limit of 45 minutes plus 500 mg Amoxicillin and 250 mg Metronidazole (AM) prescribed on the day of treatment, every 8 hours for 7 days.
  Interventions: Procedure: One-Stage Full Mouth Debridement; Drug: Amoxicillin 500mg; Drug: Metronidazole 400mg

INTERVENTIONS:
Procedure: One-Stage Full Mouth Debridement — Periodontal debridement
Drug: Amoxicillin 500mg — Administration of Amoxicillin 500mg prescribed on the day of treatment tid for 7 days.
  Arms: FMUD + AM
Drug: Metronidazole 400mg — Administration of Metronidazole 400mg prescribed on the day of treatment tid for 7 days.
  Arms: FMUD + AM
Drug: Amoxicillin Placebo — Administration of Placebo on the day of treatment tid for 7 days.
  Arms: FMUD + Placebos
Drug: Metronidazole Placebo — Administration of Placebo on the day of treatment tid for 7 days.
  Arms: FMUD + Placebos

SUMMARY:
Periodontitis is an inflammatory disease characterized by a dysbiotic microbiome which can lead to bone destruction and tooth loss. Several studies had been reported the association to periodontal disease with systemic conditions and this relation suggests and axis that links oral and gut microbiome. In order to clarify the impact of periodontal condition on gut microbiome, we aim to evaluate the clinical, immunological parameters and the microbiological condition by sequencing of subgingival biofilm and stool samples both before and after non-surgical periodontal treatment with and without antibiotics as adjunct.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage III/IV and grade C Periodontitis
* Presence of at least 20 teeth
* Good general health

Exclusion Criteria:

* Pregnant or lactating
* Were suffering from any other systemic diseases (e.g., cardiovascular, diabetes)
* Received antimicrobials in the previous 6 months
* Received a course of periodontal treatment within the last 6 months
* Were taking long-term anti-inflammatory drugs
* Smoking habits

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change in the oral-gut axis microbiome at 3 months | Baseline and 90 days
  Concentration of bacteria in the subgingival biofilm and stool samples

SECONDARY OUTCOMES:
Change of biofilm gene expression on oral microbiome at 3 months | Baseline and 90 days
  RNA-seq of 3 samples FMUD+AM group and validation by quantitative polymerase chain reaction
Change of the baseline inflammatory markers levels in gingival crevicular fluid (pg/uL) and stool samples | Baseline and 90 days
  Concentration of cytokines and biomarkers in gingival crevicular fluid and in stool samples
Change of the baseline relative clinical attachment level at 3 months | Baseline, 30 days and 90 days
  Distance from the bottom of the pocket to the stent margin.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, UNICAMP, Piracicaba, São Paulo, Brazil